CLINICAL TRIAL: NCT06142292
Title: Mitigating Mental and Social Health Outcomes of COVID-19: a Counseling Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Idaho State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2024-98; NCT05739526 (obsolete NCT alias)
Record Dates: First submitted 2023-11-17; First posted 2023-11-21 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-07

CONDITIONS: Social Determinants of Health; Mental Health Issue; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clients (Experimental): All participants will be asked to complete the following:
  participate in 12 individual mental health counseling sessions participate in 3 group counseling sessions
  Interventions: Behavioral: Individual counseling; Behavioral: Group counseling

INTERVENTIONS:
Behavioral: Individual counseling — Individual counseling sessions with a licensed mental health counselor
Behavioral: Group counseling — Group counseling sessions with a licensed mental health counselor

SUMMARY:
The goal of this clinical trial is to develop a comprehensive mental health counseling program purposed to address the social determinant of health impacts of the coronavirus disease of 2019 (COVID-19). The main questions the investigators aim to answer are: 1) What are the mental and social determinant of health impacts of a COVID-19 diagnosis, and 2) What are the impacts of a counseling program implemented to address those impacts? Participants will participate in individual interviews, attend individual and group counseling, and be provided resources related to their social determinants of health needs.

DETAILED DESCRIPTION:
The social determinants of health (SDOH) are an important social justice issue affecting various quality of life outcomes (e.g., physical and mental health). COVID-19 has disproportionately affected the SDOH of underserved and minority communities, including those in New Mexico (NM) and Idaho (ID). However, there is a lack of research on specifically how COVID-19 has affected individuals' SDOH, inhibiting prevention and response from mental health professionals and their interprofessional collaborators. Counselor education researchers have also not yet conducted outcome-based studies in this area. This research will support the development of a comprehensive, SDOH-focused mental health counseling program aimed to assess for and address the SDOH impacts of COVID-19 for individuals in NM and ID. This research will include in-depth assessment of participants' SDOH needs pertinent to COVID-19. Counseling may cover topics directly related, but also adjacent, to the participants' COVID-19 diagnosis and its impact. Participants will be provided resources and referrals specific to those needs, and engage in individual and group mental health counseling services aimed to mitigate the adverse mental and social health outcomes of COVID-19. Thus, this research should provide understanding of (1) the SDOH impacts of COVID-19, (2) feasibility of a mental health counseling program purposed to address such needs, and (3) the mental health and SDOH-related impacts of such a counseling program.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* tested positive for COVID-19 at some point in time
* reports experiencing economic, social, educational, healthcare, and/or environmentally related challenges due to their COVID-19 diagnosis
* is not currently receiving mental health counseling services
* resides in the State of New Mexico (NM) or the State of Idaho (ID)
* has access to the internet (not necessary for counseling services, but to complete interviews/assessments)
* has not experienced active suicidal or homicidal ideation or active psychosis in the last six months

Exclusion Criteria:

* is not at least 18 years of age
* has not received a COVID-19 diagnosis within the last year
* does not report experiencing economic, social, educational, healthcare, and/or environmentally related challenges due to their COVID-19 diagnosis
* is currently receiving mental health counseling services
* does not have access to the internet
* has experienced active suicidal or homicidal ideation or active psychosis in the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Social and Mental Health Outcomes of COVID-19 | Up to three weeks
  Semi-structured, audio recorded interview to gather information on the SDOH and mental health impacts of COVID-19
Social determinants of health challenges | Up to three weeks
  Self-report measure of SDOH needs through the WellRx (Page-Reeves et al., 2016)
Changes in mental health | Pre/post individual sessions (approx. 12 weeks)
  Self-report quantitative measures of depression, anxiety, and wellness
Program Feasibility/Impact | At end of study/approx. 12 weeks
  Qualitative data collected via semi-structured exit interviews of participants and their counselors
Recruitment and retention data | Throughout study, monthly
  To understand the feasibility of this study, the investigator will note how many individuals were recruited for the study (Months 1 and 2), the number of individuals who consent to participate (Months 1 and 2), and then in subsequent months, the investigator will note the number of participants who remain in the study. Each month, the investigator will also make note of how many self-report measures each participant completes on a monthly basis.

CONTACTS AND LOCATIONS:
Locations (1):
- Idaho State University, Meridian, Idaho, United States

IPD SHARING:
Plan to Share IPD: No